CLINICAL TRIAL: NCT03140501
Title: Improving Self-Management Skills Among People With Spinal Cord Injury
Acronym: MobileApp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Ben Mortenson, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 440872
Record Dates: First submitted 2017-04-26; First posted 2017-05-04 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Spinal Cord Injuries; Self-Management; Mobile Application
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Mixed-methods, rater-blinded, randomized controlled trial with a stepped wedge design (i.e., delayed intervention control group). The qualitative portion will consist of semi-structured interviews with a sub-sample of the participants.
Who Masked: Outcomes Assessor
Masking Description: Since it is not possible to blind the participants or the interventionists, a single blind study design will be employed in which data collectors are blinded to participants' group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): Participants randomized to this group will receive the intervention, the mobile application ("app"), immediately after baseline data are collected.
  Interventions: Device: Mobile application ("app")
- Delayed intervention (Other): Participants randomized to this group will receive the intervention, the mobile application ("app"), after a three month delay.
  Interventions: Device: Mobile application ("app")

INTERVENTIONS:
Device: Mobile application ("app") — The self-management app has 3 main features: 1) SCI-specific education modules; 2) a "circle-of-care" in which the users select health allies (formal and informal caregivers); and 3) a variety of tools to assist with goal identification, symptom/behaviour tracking, etc. The intervention will involve 5-6 contacts that occur over a 3-month period and ongoing use of the app. There will be 1 to 2 in-person sessions, where the principles of self-management are reviewed, self-management goals are identified, and features of the app are explained. Over the next month, there will be 2 follow-up contacts to review any questions/issues participants have. Participants can set additional goals during this time. Over the last 2 months, there will be monthly contacts to address the same issues.

SUMMARY:
The goal of our study is to evaluate the use of a self-management application ("app") that the investigators have developed to help facilitate self-management among individuals with SCI who live in the community. The main purpose is to create and fulfill individual self-management goals. Other purposes include improving self-management and health conditions related to SCI.

During the initial phase, participants (SCI clinicians and patients with SCI) reported positive usage of the self-management app and all agreed it would benefit people with SCI. With the widespread use of portable electronic devices, an opportunity exists to help patients and informal caregivers on the journey from rehabilitation to integration back into the community. The investigators will use a randomized controlled trial (randomly putting participants into two groups), including both surveys and interviews. The study will involve the use of the app that focuses on the self-management of SCI, along with five to six in-person or telephone meetings over a three-month period.

Our proposal is original in that it will be one of the few randomized control trials for e-health interventions for self-care management for those with SCI. The overall goals of the study is to develop an affordable self-management app that can be used to encourage self-management in people living with SCI. This app would be used along with other health problem specific apps that are more detailed and expensive, while helping participants to manage their long-term health problems related to their SCI in an easily usable and affordable form.

DETAILED DESCRIPTION:
Most people with spinal cord injury (SCI) will develop debilitating secondary conditions, such as autonomic dysreflexia and pressure ulcers. Self-management programs, which recognize patients' central role in managing their condition, have been found to improve health-outcomes in a variety of populations, such as those living with diabetes and asthma. Given the increase in health care costs and funding constraints, alternative self-management interventions are being explored, such as the use of electronic health (e-health) treatments. Despite the potential benefits of self-management among people with SCI, the investigators were able to identify little experimental research in this area.

Our goal is to evaluate the efficacy of a broad-based self-management application ("app") the investigators have developed to facilitate the improvement of self-management skills among community-dwelling individuals with SCI. The primary outcome is attainment of self-selected self-management goals. Secondary outcomes include general and self-management self-efficacy, secondary conditions related to SCI, self-reported healthcare utilization, self-reported health events, and app usage data.

During the preliminary phase of the study, participants (SCI clinicians and patients with SCI) reported favourable usage of the self-management app and unanimously agreed it would benefit people with SCI. With the ubiquity of portable electronic devices, an opportunity exists to help participants and informal caregivers navigate the journey from rehabilitation to integration back into the community. The research team will use both quantitative and qualitative methods involving a rater-blinded, randomized controlled trial with a stepped wedge design and semi-structured interviews. The participant-specific intervention will involve the use of the self-management app focusing on the self-management of SCI accompanied by five to six in-person or telephone/Skype contacts that will occur over a three-month period.

Our proposal is original in that it will be one of the few randomized controlled trials in the area of e-health interventions for self-care management for those with SCI. Although the use of qualitative and qualitative methods has been recommended in randomized controlled trials, relatively few studies have used this design, so the proposed study may provide a model for assessing the effectiveness of other self-management interventions. The overall purpose of the study is to develop an effective self-management application that can be used to promote self-management in a variety of populations and is less resource intensive. This app would be complementary to other complication specific apps that are more in-depth and expensive to deliver, while providing an accessible and affordable form of tertiary prevention for those who develop secondary complications.

ELIGIBILITY:
Inclusion Criteria:

* Have been discharged from inpatient rehabilitation following a spinal cord injury at least one year prior
* Are living in the community setting
* Are 19 years of age or over
* Speak, read, and write English
* Have reliable access to internet
* Are capable of providing your own informed consent

Exclusion Criteria:

* Are unable to provide informed consent (due to severe mental illness or traumatic brain injury)
* Have previously used a self-management mobile app focused on spinal cord injury (including SCI Health Storylines)
* Have cognitive impairments that impact memory, communication or ability to complete questionnaires.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scaling (GAS) | At 0 months (baseline), 3 months after baseline, 6 months after baseline, and 9 months after baseline
  GAS is a promising approach for evaluating psychosocial interventions in community settings. This measure will be used to identify self-management goals that participants want to achieve. Objective outcomes are identified that indicate degrees of attainment of participant-selected goals on a five-point scale ranging from -2 to +2, where -2 is a much worse than expected outcome, 0 represents attaining the goal (the anticipated outcome) and 2 means a much better than expected outcome, and then aggregate T-scores are calculated. The minimally clinically important change for GAS is 10, based on the linear T-score, which represents a change in score from the anticipated values.

SECONDARY OUTCOMES:
Self-Efficacy for Managing Chronic Disease Scale | At 0 months (baseline), 3 months after baseline, 6 months after baseline, and 9 months after baseline
  This scale is designed to evaluate confidence in managing long-term disease. It has been used extensively in many different populations including people with spinal cord injury to evaluate self-management interventions. Each of the 6-items are rated on a scale of 1-10 (with 1 indicating 'not at all confident' and 10 indicating 'totally confident') and an average score is calculated.
Spinal Cord Injury Secondary Conditions Scale | At 0 months (baseline), 3 months after baseline, 6 months after baseline, and 9 months after baseline
  This is one of two outcome measures that assesses self-efficacy. This scale targets secondary conditions related to spinal cord injury that have both direct and indirect impacts on health. The 16-item scale uses a 4-point ordinal scale ranging from 'no problem' to 'significant problem' with the total score ranging from 0-49.
Self-Reported Healthcare Utilization | Throughout the study, up until the end-point (9 months)
  Healthcare utilization will be measured by having participants record visits to see a physician, visits to hospital emergency departments, number of hospitalizations, and the number of nights spent in hospital. Although there may be recall issues within self-reported healthcare utilization, it has been found to be highly correlated with days in hospital (r=0.83) (17). Participants will complete a weekly journal to help improve the accuracy of the report.
Spinal Cord Independence Measure III | At 0 months (baseline)
  This is a disability scale developed to specifically address the ability of spinal cord injury patients to perform basic activities of daily living independently. It assesses three areas: 1) self-care (e.g., feeding, grooming, bathing, and dressing), 2) respiration and sphincter management, and 3) mobility (bed and transfers and indoor/outdoor). The item scores are weighted related to the assumed clinical relevance.
American Spinal Injury Association Impairment Scale | At 0 months (baseline)
  This is a clinical examination conducted to test whether sensation is 0-absent; 1-impaired; or 2-normal. Muscle function is rated from 0-total paralysis to 5-normal (active movement, full range of motion against significant resistance). Although the investigators will be unable to administer the measure as it requires significant and specialized training, a research team member will ask participants if they have been evaluated and what their motor and sensory impairment level is, if they know. This is included in the demographics form.
Interpersonal Support Evaluation List (ISEL) | At 0 months (baseline), 3 months after baseline, 6 months after baseline, and 9 months after baseline
  This list measures the perceptions of social support among individuals in the general population. It examines the ways in which others affect persons' responses to stressful events. It consists of a list of 40 statements concerning the perceived availability of potential social resources. The items are counterbalanced for desirability - half the items are positive statements about social relationships while the other half are negative statements. Items fall into four 10-item sub-scales: tangible support, appraisal support, self-esteem support, belonging support.
Technology Readiness Index | At 0 months (baseline)
  This is a multiple-item scale that measures an individual's readiness to embrace new technologies.
Leisure Time Physical Activity Questionnaire-SCI | At 0 months (baseline), 3 months after baseline, 6 months after baseline, and 9 months after baseline
  This is an SCI-specific, self-report measure of leisure time physical activity (LTPA) that assesses minutes of mild, moderate, and heavy intensity LTPA performed over the previous 7 days. It is unique because it captures different types of LTPA performed at different intensities.
Health Care Climate Questionnaire | At 0 months (baseline), 3 months after baseline, 6 months after baseline, and 9 months after baseline
  This measure is used to access patients' perceptions of the degree to which their specific doctor is autonomy supportive, and it can be used to assess patients' perceptions of the degree to which their team of health care providers is autonomy supportive.
Amount of informal/formal caregiving | At 0 months (baseline), 3 months after baseline, 6 months after baseline, and 9 months after baseline
  This measure is used to determine the amount of caregiving that participants require from their formal and informal caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Ben Mortenson, PhD, Principal Investigator — University of British Columbia
Locations (1):
- GF Strong Rehabilitation Center, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mortenson WB, Mills PB, Adams J, Singh G, MacGillivray M, Sawatzky B. Improving Self-Management Skills Among People With Spinal Cord Injury: Protocol for a Mixed-Methods Study. JMIR Res Protoc. 2018 Nov 14;7(11):e11069. doi: 10.2196/11069. PMID 30429114